CLINICAL TRIAL: NCT02482948
Title: "Prospective, Randomized, Multi-Center, Efficacy Non-inferiority Study of MEDIHONEY® Gel Versus Collagenase for Wound Debridement"
Brief Title: MEDIHONEY® Gel Versus Collagenase for Wound Debridement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Derma-MH001
Record Dates: First submitted 2015-06-12; First posted 2015-06-26 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Ulcer; Wounds
Keywords: Debridement; collagenase; leptospermum honey
MeSH Terms: conditions — Ulcer; Wounds and Injuries | interventions — Collagenases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collagenase (Active Comparator): This is an enzymatic debridement agent to remove non-viable tissue from wounds to be applied daily
  Interventions: Drug: Collagenase
- Active leptospermum honey (Active Comparator): This is an active medicinal grade honey used to promote autolytic debridement and applied daily
  Interventions: Device: Active Leptospermum Honey (Medihoney)

INTERVENTIONS:
Device: Active Leptospermum Honey (Medihoney) — STudy agent to be applied to the wound daily.
  Other Names: Medihoney
  Arms: Active leptospermum honey
Drug: Collagenase — Study agent to be applied daily to the wound.
  Other Names: Santyl
  Arms: Collagenase

SUMMARY:
The purpose of this study is to compare how well two products, Active Leptospermum Honey (ALH) (MEDIHONEY® Gel) and Collagenase (Santyl®), in removing the nonviable (non living) tissue.

DETAILED DESCRIPTION:
BACKGROUND

An important aspect of wound bed preparation for healing or grafting is the recognition that wounds often have underlying pathogenic abnormalities that cause necrotic tissue to accumulate. Therefore, in order to facilitate wound progression, repeated removal of necrotic tissue may be necessary as long as the wound is chronic. Debridement is defined as the removal of nonviable material, foreign bodies, and poorly healing tissue from a wound. Although surgeons recognize the importance of debridement, few data have been generated in randomized trials to support its use. Traditionally, debridement has been undertaken as a single therapeutic step within defined time frames. The most direct form of debridement is surgical excision. Although this may be applicable for acute wounds, it is unlikely to remove the necrotic burden that may continually accumulate in a chronic wound. Although there are other forms of debridement including enzymatic and biologic; in the case of non-healing wounds, the form of debridement with the most compelling evidence of healing efficacy is autolytic debridement , Therefore, for patients who are poor candidates for surgical debridement or have limited access to a surgeon, autolytic debridement may be considered an effective form of continuous debridement.

2.1 Primary Objective

The primary objective of this study is to evaluate the non-inferiority of MEDIHONEY® Gel (Active Leptospermum Honey-ALH Gel) compared to (Santyl) Collagenase, two FDA cleared/approved treatments, with respect to the percent reduction of necrotic (including slough and eschar) tissue in the wound at the end of 14 days +/- 2 days.

2.2 Secondary Objective

The secondary objective of this study is to compare the two treatment groups with respect to the percent reduction from randomization for necrotic tissue (including slough and eschar) at weeks 1, 3 and 4 +/- 2 days.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent has been obtained from the subject.
* Subject is able and willing to comply with study procedures.
* Subject is able to comply with weekly visits.
* Subject is 18 years of age or older.
* There is presence of at least 50% or greater necrotic tissue (including slough and eschar) in the wound bed and a total wound surface area of > 1cm2 to < 64cm2.
* Subject will not have currently used parenteral or oral antibiotics except for UTI.
* Diabetic subjects: HbA1c < 12.0 % within 90 days preceding enrollment.
* Pre-albumin greater than 16 mg/dl within 90 days preceding enrollment.
* Subject with a pressure ulcer must be currently receiving adequate pressure redistribution to the affected area via group 2 or 3 specialty bed, a static wheel chair cushion while patient is out of bed.
* Subject with diabetic plantar surface ulcer will use an offloading boot if ambulatory.
* Subject with a venous ulcer must be currently receiving and using compression therapy that can be managed daily.
* Subject and caregiver are trainable and able to perform dressing changes.
* Subject has no allergies to collagenase or honey.
* Subject has no allergies to semi-occlusive or absorptive secondary dressing.
* If subject has multiple wounds only the wound that fits the inclusion criteria will be selected. If more than one wound meets criteria then the largest wound will be selected.

Exclusion Criteria:

* Steroid use >5mg daily.
* Subject is unable to cooperate with offloading and/or compression recommendations.
* ABI = or >0.8 if the wound is located on a lower extremity.
* Wound has the presence of callus requiring sharp or surgical debridement within 3 days prior to randomization and/or needs debridement using any method other than the study agent throughout study treatment.
* Subject has medical instability as deemed by the investigator.
* Subject is pregnant.
* Subject has participated in another clinical trial or wound dressing evaluation in the 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Necrotic tissue reduction | two weeks
  Necrotic tissue percent reduction in the wound at the end of 14 days

SECONDARY OUTCOMES:
Percent wound reduction | 4 weeks
  Percent wound reduction from randomization at weeks 1, 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Patel, MD, Principal Investigator — Innovative Healing Systems
Locations (1):
- Innovative Healing Systems, Tampa, Florida, United States